CLINICAL TRIAL: NCT04062162
Title: Is the Walking Football a Feasible Approach to Improve Health-related Quality of Life in Men With Prostate Cancer Receiving Androgen Deprivation Therapy? the PROSTATA_MOVE Randomized Controlled Trial.
Brief Title: Walking Football as a Supportive Medicine for Patients With Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Associacao de Investigacao de Cuidados de Suporte em Oncologia (Other)
Collaborators: Centro Hospitalar de Vila Nova de Gaia/Espinho, E.P.E. (Other Government); University of Beira Interior (Other); Federação Portuguesa de Futebol (Unknown); University Institute of Maia (Other); Câmara Municipal de Gaia (Unknown)
Responsible Party: Principal Investigator, Andreia Capela, Medical oncologist at Centro Hospitalar de Vila Nova de Gaia/Espinho, E.P.E., Associacao de Investigacao de Cuidados de Suporte em Oncologia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AICSO
Record Dates: First submitted 2019-08-08; First posted 2019-08-20 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Prostate Cancer; Androgen Deprivation Therapy
Keywords: Prostate Cancer; Androgen Deprivation Therapy; Walking football
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Active Comparator): Walking football training
  Interventions: Behavioral: Walking football training
- Control group (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Walking football training — Intervention will involve 3 sessions per week of a structured and supervised walking football program over 16 weeks. Each session will include a warm-up, followed by the practice of specific exercises where specific technical skills (pass, dribble, shot), motor skills (agility, coordination, balance) and physical fitness (cardiorespiratory and musculoskeletal capacity) will be enhanced, ending with a structured game (7x7) of walking football and a cooldown.
  Other Names: Exercise training
  Arms: Interventional group

SUMMARY:
Androgen deprivation therapy (ADT) is widely used in men with prostate cancer (PCa) to delay disease progression and enhance survival. The use of ADT is often associated with a vast spectrum of side effects that considerably reduce quality of life. Exercise has been proposed as a non-pharmacological strategy to counter some adverse effects of ADT among patients with PCa. Particularly, recreational football-based interventions have been suggested as an enjoyment approach to involve patients with PCa in regular exercise practice. Given its intermittent nature and vigorous efforts, adverse events associated with recreational football practice have been reported. To handle this issue and to involve patients with PCa in recreational football practice, walking football has emerged as a more suitable exercise modality

DETAILED DESCRIPTION:
This study was design as a randomized controlled trial, with two study arms, which aims to analyse the feasibility, safety of a supervised walking football program in patients with PCa. Moreover, the effects on health-related quality of life; bone mineral density; body composition; physical fitness; physical activity levels; inflammatory and metabolic profile; cognitive function; and cost-effectiveness will be complementarily analysed.

Recruitment will be conducted by invitation of Centro Hospitalar de Vila Nova de Gaia/Espinho (CHVNG/E; Vila Nova de Gaia, Portugal, E.P.E) oncologists and urologists. Patients who agree to participate in this study will be referred to a study coordinator (medical oncologist) and will be randomly allocated (1:1 ratio) to one of the two study-arms.

In addition to standard PCa care, patients in the interventional group (IG) will perform 3 times per week a supervised Walking Football Program over 16 weeks and plus 16 additional weeks.

Patients allocated to control group (CG) will receive standard PCa medical care and will be instructed to maintain daily-life routines. After the first 16 weeks, the control group patients' will be invited to join and preform the exercise intervention (additional 16 weeks).

Walking football exercise sessions will be conducted on an indoor sports hall, supervised by one exercise physiologist and a football coach. Exercise intensity will be monitored through heart rate and rated perceived exertion.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with PCa
* Under castration therapy for more than 3 months
* Planned to be under castration for more than 6 months
* Follow-up at the Medical Oncology department and/or Urology department of the Hospital Center Vila Nova de Gaia/Espinho.

Exclusion Criteria:

* Medical or surgical contraindications for exercise.
* T-score < -2.5

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 50 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate. | Baseline
  Assessed by the number of enrolled patients divided by the number of invited patients.
Withdrawal rate | Change from baseline to 32 weeks
  Assessed by the number of withdrawal patients
Appropriateness of outcomes assessments. | Change from baseline to 32 weeks
  Assessed by the percentage of completed data.
Adherence to intervention. | Change from baseline to 32 weeks
  Assessed by the number of completed sessions and the number of missed sessions.
Rate of Enjoyment | Change from baseline to 32 weeks
  Assessed by the self-reported exercise sessions' enjoyment using a likert scale (1 [lowest] to 5 [highest] points).
Health-related quality of life | Change from baseline to 32 weeks
  Using EORTC PR25, EQ-5D-5L and SF-6D questionnaire.

SECONDARY OUTCOMES:
Bone Mineral Density | Change from baseline to 32 weeks
  Assessed by a whole-body dual-energy X-ray absorptiometry (DXA) scan.
Body composition | Change from baseline to 32 weeks
  Assessed by a whole-body dual-energy X-ray absorptiometry (DXA) scan.
Aerobic capacity | Change from baseline to 32 weeks
  Assessed by a symptom-limited exercise test on a treadmill
Maximal isometric handgrip strength | Change from baseline to 32 weeks
  Assessed using a digital handgrip dynamometer.
Maximal isometric lower limb strength | Change from baseline to 32 weeks
  Assessed using a digital handgrip dynamometer.
Lower limb functionality | Change from baseline to 32 weeks
  Assessed by the 30-seconds sit-to-stand test
Static balance | Change from baseline to 32 weeks
  Assessed by the single leg stance test
Habitual physical activity levels | Change from baseline to 32 weeks
  Assessed using accelerometers
Exercise intensity - External load | Change from baseline to 32 weeks
  Distance (km) assessed using GPS tracking during exercise
Exercise intensity - Internal load | Change from baseline to 32 weeks
  Assessed by the heart rate
Exercise intensity - Rating of perceived exertion | Change from baseline to 32 weeks
  Assessed using a 6-20 borg scale (minimum effort = 6; maximum effort = 10).
Cogntive function | Change from baseline to 32 weeks
  Assessed by the Montreal Cognitive Assessment
Blood pressure | Change from baseline to 32 weeks
  Assessed using a digital sphygmomanometer
Resting heart rate | Change from baseline to 32 weeks
  Assessed using a digital sphygmomanometer
LDL-cholesterol | Change from baseline to 32 weeks
  Blood sample will be taken for analysis of levels of LDL-cholesterol
HDL-cholesterol | Change from baseline to 32 weeks
  Blood sample will be taken for analysis of levels of HDL-cholesterol
Total cholesterol | Change from baseline to 32 weeks
  Blood sample will be taken for analysis of levels of total cholesterol
Triglycerides | Change from baseline to 32 weeks
  Blood sample will be taken for analysis of levels of triglycerides
Prostate specific antigen (PSA) | Change from baseline to 32 weeks
  Blood sample will be taken for analysis of levels of PSA
Creatinine | Change from baseline to 32 weeks
  Blood sample will be taken for analysis of levels of creatinine
High sensitivity C-reactive protein (HS-CRP) | Change from baseline to 32 weeks
  Blood sample will be taken for analysis of levels of HS-CRP
N-terminal type B natriuretic peptide (NT-proBNP) | Change from baseline to 32 weeks
  Blood sample will be taken for analysis of levels of NT-proBNP
Vitamin D | Change from baseline to 32 weeks
  Blood sample will be taken for analysis of levels of vitamin D
Osteocalcin | Change from baseline to 32 weeks
  Blood sample will be taken for analysis of levels of
C-Telopeptide of Collagen Cross-links (CTx) | Change from baseline to 32 weeks
  Blood sample will be taken for analysis of levels of CTx
Bone Specific Alkaline Phosphatase (BSAP) | Change from baseline to 32 weeks
  Blood sample will be taken for analysis of levels of BSAP
Tartrate-Resistant Acid Phosphatase (TRAP) | Change from baseline to 32 weeks
  Blood sample will be taken for analysis of levels of TRAP
Glycated hemoglobin | Change from baseline to 32 weeks
  Blood sample will be taken for analysis of levels of glycated hemoglobin
Testosterone | Change from baseline to 32 weeks
  Blood sample will be taken for analysis of levels of testosterone

CONTACTS AND LOCATIONS:
Overall Officials: Andreia Capela, MD, Principal Investigator — Centro Hospitalar Vila Nova de Gaia / Espinho, EPE
Locations (1):
- Centro Hospitalar Vila Nova de Gaia / Espinho, Vila Nova de Gaia, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Capela A, Antunes P, Coelho CA, Garcia CL, Custodio S, Amorim R, Costa T, Vilela E, Teixeira M, Amarelo A, Silva J, Joaquim A, Viamonte S, Brito J, Alves AJ. Effects of walking football on adherence, safety, quality of life and physical fitness in patients with prostate cancer: Findings from the PROSTATA_MOVE randomized controlled trial. Front Oncol. 2023 Mar 21;13:1129028. doi: 10.3389/fonc.2023.1129028. eCollection 2023. PMID 37025594